CLINICAL TRIAL: NCT02104037
Title: Liraglutide in Spinal Fluid
Acronym: LIRA-CSV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mikkel Christensen (Other)
Responsible Party: Sponsor-Investigator, Mikkel Christensen, Dr., University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-2-2011-027
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Liraglutide Blood-brain Transfer
MeSH Terms: interventions — Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Liraglutide treated patients (Experimental)
  Interventions: Procedure: Lumbar puncture

INTERVENTIONS:
Procedure: Lumbar puncture

SUMMARY:
The purpose of this study is to investigate transfer of liraglutide from blood to cerebrospinal fluid.

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabetes treated with liraglutide 1.8 mg for 1 month and 5% weight loss

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
cerebrospinal fluid concentration of liraglutide | time 60 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetes Research Division, Department of Medicine, Hellerup, Denmark